CLINICAL TRIAL: NCT01278810
Title: A Phase I ,Single Center, Open-labeling, Single and Dose-escalating Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of Oral Novel ERa36 Modifier Icaritin in Advanced Breast Patients
Brief Title: Phase I Study of Novel Estrogen Receptor(ER) a36 Modifier Icaritin in Advanced Breast Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Shenogen Biomedical Co., Ltd (Industry)
Responsible Party: xubinghe, Cancer institute & hospital, chinese academy of medical sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG0929ICR
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2010-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Icaritin,; ERa36
MeSH Terms: conditions — Breast Neoplasms | interventions — icaritin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Icaritin (Experimental)
  Interventions: Drug: Icaritin

INTERVENTIONS:
Drug: Icaritin — 50mg,100mg,200mg,300mg,400mg,500mg ascending-multiple oral dose, Qd, single dose and continuing dose 28 days, to assess the safety,tolerance and pharmacokinetics of icaritin
  Other Names: IC-162

SUMMARY:
To assess safety, tolerance and PK profile of different doses(50mg,100mg,200mg,300mg, 400mg, 500mg,QD)of Icaritin in advanced breast cancer Patients in China

DETAILED DESCRIPTION:
ERa36 predominantly localizes on the plasma membrane and in the cytoplasm and mediates a membrane-initiated "nongenomic" signaling pathway. Membrane-initiated estrogen signaling has been linked to rapid responses to estrogen and generally activates signaling pathways like MAPK/ERK, phosphatidylinositol-3-kinase, and protein kinase C pathways. Preclinical study demonstrated that ERa36 was expressed in tumor cells and might be the driving force of breast cancer cell proliferation. 40% of breast cancer tumors which used to be considered as ER negative also express ERa36. In the former study the investigators found that 40% of ERa66-positive breast cancer patients express high levels of ERa36 in their tumors, and this subset of patients are less likely to benefit from tamoxifen treatment compared with those with ERa66-positive/ERa36-negative tumors.

Icaritin is a newly discovered small molecular compound which is high selective ERa36 modulators and perhaps will be a very promising new drug to treat advanced breast cancer by targeting this nongenomic pathway. It was showed that it can inhibit the growth of breast cancer cells both in vitro and in vivo. The investigators have completed the preclinical PK&PD and toxicity studies in animals and now move on to test it in a FIM clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age ≥ 18 years old and ≤ 65 years old
2. The patients with advanced breast tumors who are confirmed through histologic or cytologic diagnosis with ER positive or investigator think that subjects will benefit from the trial
3. The advanced breast cancer patients which relapse or failure from previous standard treatment
4. 19 ≤ BMI index ≤ 30
5. No serious heart, liver,lung and kidney diseases
6. Received at least once anti-cancer treatment (including chemotherapy, radiotherapy, biological or endocrine treatment). And the last treatment must be at least four weeks before study enrollment or more than 5 times half life. The surgery treatment must be more than three months
7. Life expectancy of at least 12 weeks
8. Patients which can cooperate to observe AE and efficacy
9. No any other concurrent anti-cancer treatment
10. A signed informed consent must be obtained prior to performing any study specific procedures
11. ECOG Performance Status of 0,1
12. Female:Women with childbearing potential must have a negative pregnancy test performed

Exclusion Criteria:

1. Have a known hypersensitivity to flavonoid drugs
2. Hepatic:

   * ALB >limit if normal
   * TB> the upper limit of normal
   * ALT and AST > upper limit of Normal

   Renal:
   * Serum Creatinine > 1.5 times the upper limit of normal

   Bone marrow:
   * Absolute neutrophil count (ANC) < 1.5 × 109/L
   * Platelet count < 90 × 109/L
   * Hemoglobin < 9 g/dL
3. PT/APTT > 1.25 times the upper limit of normal
4. Suffered from thrombotic disease
5. Serum Ca > the upper limit of normal
6. Not recovered from toxic effects of previous anti-cancer treatments or surgery
7. Any serious or uncontrollable concomitant systemic disorder (such as unstable respiratory disorders, cardiovascular, hepatic or kidney disorders.) or active infection which will influence the clinical trial
8. CNS metastases or invade requiring treatment for unstable status or various psychiatric disorders
9. No malabsorption or other disease which will affect the drug absorption,distribution,metabolism and excretion
10. Concurrent other malignancies with the exception of cervical cancer in situ or squamous Cell Carcinoma of the Skin

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To assess safety of icaritin in breast cancer patients | 1-2 YEAR
  to find the dose-limiting toxicity(DLT)and maximal tolerated dose(MTD)of icaritin in breast cancer patients

SECONDARY OUTCOMES:
To assess pharmacokinetic profile of icaritin in breast cancer patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Binghe Xu, MD, Principal Investigator — Cancer institute & hospital
Locations (1):
- Cancer institute & hospital, chinese academy of medical sciences, Beijing, Beijing Municipality, China